CLINICAL TRIAL: NCT01222988
Title: Improving Maintenance Following Very Low Calorie Diet: The Sustain Lost Weight (SLW) Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Gretchen E. Ames, Ph.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-002960
Record Dates: First submitted 2010-10-12; First posted 2010-10-18 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- very low calorie diet program (Other)
  Interventions: Dietary Supplement: Optifast Products

INTERVENTIONS:
Dietary Supplement: Optifast Products — Optional Optifast products offered once every other week X 6 months; then monthly.
  Other Names: Optifast Dietary Supplements

SUMMARY:
Obtain a preliminary assessment of the feasibility and acceptability of delivering the sustained lost weight (SLW) intervention in a real-world clinical setting for patients who have completed a 21-week very low calorie diet (VLCD).

Hypothesis: Intervention will be feasible to implement as evidenced by the ability to recruit and retain participants and acceptable to participants as evidenced by self-report of satisfaction with the program and adoption of weight maintenance behaviors.

Secondary Aim: Obtain a preliminary assessment of the effectiveness of the sustained lost weight (SLW) intervention for patients who have completed 21 weeks of a very low calorie diet (VLCD).

Hypothesis: Greater than 75% of participants who receive this novel approach, where maintenance behaviors are individualized based on resting metabolic rate and a physical activity factor, will regain greater or equal to 10 kg. at week 52 follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Completed fast and transition period of the OPTIFAST® program
* Be able to participate fully in all aspects of the study
* Willing to refrain from participating in additional weight loss interventions for the duration of the study
* Willing to provide written informed consent.

Exclusion Criteria:

* Myocardial infarction within 6 months
* Unstable angina
* Stroke
* Chronic steroid use
* Active peptic ulcer disease
* Advanced cirrhosis
* Active hepatitis
* Advanced renal disease
* Active thrombophlebitis
* Recent skeletal fractures
* Use of lithium
* Pancreatitis
* Pregnancy
* Type 1 diabetes mellitus
* History of diabetic ketoacidosis
* Active bulimia nervosa
* Severe depression
* Psychosis
* Substance abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Treatment Feasibility | 52 weeks
  Treatment will be considered feasible if greater than 50 % of participants attend a minimum of 17 of 20 sessions. The treatment will be considered acceptable for further study if greater than 50% of participants rate the maintenance program with a mean score of 6 or higher.

SECONDARY OUTCOMES:
Weight Gain Analysis | 52 weeks
  Weight regain from week 1 to 52 will be analyzed. Patients who discontinue the study or are lost to follow-up will be assumed to have gained more than 10 kg at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Ames, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States